CLINICAL TRIAL: NCT02025582
Title: The Effectiveness and Efficacy of Kinesio Taping Method on Muscle Elasticity in Children Who Toe Walk
Brief Title: Kinesio Taping Effectiveness on Idiopathic Toe Walking
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hadiya Guerrero, P.T., Hadiya Guerrero, P.T., D.P.T., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-003848
Record Dates: First submitted 2013-12-27; First posted 2014-01-01 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Idiopathic Toe Walking
Keywords: idiopathic toe walking; gait disorder; gait analysis; kinesio taping; ultrasound elastography; pediatric; children; muscle stiffness; muscle elasticity
MeSH Terms: conditions — Mobility Limitation | interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kinesio tape (Experimental)
  Interventions: Device: Kinesio Tape of the Ankle

INTERVENTIONS:
Device: Kinesio Tape of the Ankle — Tibialis anterior facilitation/ gastrocnemius inhibition: Taping to be worn 3-5 days and repeated x 1
  Other Names: Kinesio Tape

SUMMARY:
Idiopathic Toe Walking (ITW) is a diagnosis normally of exclusion and likely, consequently, is approached in vastly varying ways of intervention, including serial casting, Botox injections and physical therapy. There is some evidence in the literature that children with ITW can somewhat correct their lack of heel-strike gait pattern at least temporarily. Kinesio Taping (KT) method is an intervention that is used in the outpatient physical therapy setting for various conditions such as post-operative edema, muscle facilitation of weakened rotator cuff muscles, and functional corrections in children with torticollis. This pilot study will strive to determine if KT may be effective by providing proprioceptive and neuromuscular re-education through thermal and mechanical fascial impositions, thereby improving passive joint range of motion (ROM) through reduction of passive muscle stiffness and improving ambulation through neuromuscular re-education in children with idiopathic toe walking. We will quantify passive muscle stiffness of the gastrocnemius and opposing anterior tibialis using non-invasive Shear Wave Elastography (SWE). Further we look at the kinematics and kinetics of the child's ankle during the gait cycle to further determine any effect(s) of KT on functional walking outcome measures. The intent is that the results from this study will serve as a platform from which to expound look at the long-term, if any, effects of KT on the muscle property and gait cycle pattern in children with ITW.

ELIGIBILITY:
Inclusion Criteria:

* Females and males
* 3-10 years of age
* who independently ambulate
* have a diagnosis of idiopathic toe walking

Exclusion Criteria:

* Children will be excluded if they have a diagnosis of or suspected neuromuscular disorder
* had prior treatment for ITW including bracing or including splinting in the last six months, chemodenervation, serial casting in the last six months, surgical intervention
* diagnosis of Autism or Pervasive Developmental Disorder
* history of allergic reactions to tape/adhesives.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Ankle Joint Range of Motion | At enrollment, one and two week after kinesio taping
  To evaluate effect of KT on passive ankle ROM, we will measure passive ankle ROM before and after treatment. With the child laying prone, measurements of ankle ROM will be taken using a goniometer with the knee extended and with the knee flexed at 90 degrees. The rationale for this is to differentiate gastrocnemius muscle from soleus muscle, with gastrocnemius contributing to ankle ROM loss when knee is extended because it crosses both joints.

SECONDARY OUTCOMES:
Advanced gait analysis - Change in kinetics | At enrollment, after completion of taping (2-3 weeks after enrollment)
  In children with ITW, gait changes, as measured by ankle kinetics and kinematics, have been shown as toe-walking improves. In ITW, presence of a first ankle rocker, presence of an early third ankle rocker, and predominant early ankle moment on advanced gait analysis are used to classify idiopathic toe walking into three severity groups. Changes to these parameters are used to evaluate effect of treatment on ITW. Therefore, we propose to use these parameters to classify the severity of the ITW before and after KT treatment to evaluate effect of KT on ambulation.

OTHER OUTCOMES:
Supersonic Shearwave Ultrasound Elastography: Change in muscle elasticity | At enrollment, upon completion of taping (2-3 weeks after enrollment)
  Currently, there is indirect evidence that children with ITW have increased passive stiffness of the gastrocnemius muscle, and no evidence with regard to passive stiffness of the anterior tibialis, a major ankle plantar flexion antagonist. Abnormal passive stiffness of these muscles is thought to result in the loss of passive ROM and changes to ambulation. However, direct measurements of passive muscles stiffness in children have not been able to be done, until recently. Therefore, we propose to quantify the passive muscle stiffness of the gastrocnemius muscle and anterior tibialis muscle in children with ITW before and after KT treatment using SWE.

CONTACTS AND LOCATIONS:
Overall Officials: Hadiya Guerrero, DPT, Principal Investigator — Mayo Clinic Foundation
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States